CLINICAL TRIAL: NCT04973332
Title: A Prospective, Multicenter, Randomized Controlled, Non-inferiority Study to Investigate the Effectiveness and Safety of Intracranial Embolization Stents for Endovascular Treatment of Acute Ischemic Stroke
Brief Title: Safety and Efficacy of SINOMED SR for Endovascular Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinomed Neurovita Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SINOMED SR
Record Dates: First submitted 2021-06-21; First posted 2021-07-22 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Ischemic Stroke, Acute; Brain Diseases; Cerebrovascular Disorders
MeSH Terms: conditions — Ischemic Stroke; Brain Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized controlled, non-infertility study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrombectomy-SINOMED SR (Experimental): Patients diagnosed with acute ischemic stroke within 24 hours from the onset of the stroke to the completion of femoral artery puncture, regardless of whether intravenous thrombolysis has been performed. Intracranial thrombectomy stents can be used to remove the thrombus in the large vessels of the brain in patients with ischemic stroke To restore blood flow.
  Interventions: Device: Intracranial thrombectomy stent
- Thrombectomy-Solitaire FR (Active Comparator): Intracranial thrombectomy was performed with a control product（name:Solitaire FR）
  Interventions: Device: Intracranial thrombectomy stent

INTERVENTIONS:
Device: Intracranial thrombectomy stent — Intracranial thrombectomy stents for ischemic stroke patients within 24 hours of symptom onset

SUMMARY:
A prospective, multicenter, randomized controlled, non-inferiority study to investigate the effectiveness and safety of SINOMED SR for endovascular treatment of acute ischemic stroke

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, 1:1, controlled trial with blinded outcome assessment assessing non-inferiority of SINOMED SR compared to Solitaire FR. The trial aims to randomize 220 patients 1:1 to receive SINOMED SR or Solitaire FR.The primary outcome is the Success rate of immediate recanalization.

ELIGIBILITY:
General inclusion criteria：

1. 18 years old or more;
2. NIHSS≥6 during randomization;
3. Pre-onset MRS < 2;
4. Acute ischemic stroke was diagnosed;
5. Within 24 hours from the onset of stroke to the completion of femoral artery puncture, regardless of whether intravenous thrombolysis has been performed;The time point of stroke onset was defined as the time point at which the patient's last normal condition was known;
6. The subject (or his/her guardian) agrees to participate in this study and signs the informed consent.

Image inclusion criteria：

1. When it is less than 6h (inclusive) from the onset of stroke to the completion of femoral artery puncture, patients should be examined by cranial CT or MR;
2. When it is more than 6h but less than 24h (inclusive) from the onset of stroke to the completion of femoral artery puncture, brain CT or MR should be performed and Aspects ≥6 points should be satisfied.(If immediate CT perfusion imaging or MR perfusion imaging is feasible, CTP or MRP is recommended to assist in the assessment of the infarct core, and Aspects ≥6 points shall also be satisfied);
3. DSA angiography showed acute intracranial arterial occlusion, including intracranial segment of internal carotid artery (C4-C7), middle cerebral artery (M1/M2), basilar artery and intracranial segment of vertebral artery (V4).

General exclusion criteria：

1. Neither MRI nor CT can be performed;
2. Hemorrhagic stroke or major ischemic stroke within 6 months before enrollment;
3. Severe persistent hypertension that cannot be controlled by venous hypotension, i.e., patients with SBP persistent >185mmHg and/or DBP persistent >110mmHg;
4. Suppose septic emboli or suspected bacterial endocarditis;
5. Renal failure, defined as: creatinine >3.0mg/dL(264 mol/L);
6. Blood glucose < 2.78mmol/L (50mg/dL) or >22.20mmol/L (400mg/dL);
7. decreased platelet count (< 40×109/L);
8. Known bleeding tendency, defect of coagulation factor, taking anticoagulants and INR > 3.0;
9. Pregnant or lactating women;
10. known to be severely allergic to contrast agents and known to be allergic to nickel materials;
11. The presence of diseases that may affect the assessment of neurological function (such as neurological diseases, mental diseases, etc.);
12. with heart, lung, liver function failure or other serious diseases to interventional surgery;
13. Participating in clinical trials of other drugs or devices;
14. Life expectancy less than 6 months;
15. Other conditions judged by the researcher to be unsuitable for inclusion.

Image exclusion criteria：

1. CT or MR imaging evidence of intracranial hemorrhage or known bleeding tendency;
2. CT/MR/DSA showed > occlusion (such as bilateral internal carotid artery occlusion at the same time, or anterior circulation and posterior circulation intracranial vessels occlusion at the same time, or internal carotid intracranial and extracranial segments occlusion at the same time);
3. Carotid artery dissection, carotid initial occlusion or arteritis;
4. The vascular circuitry was severe, and the intracranial thrombectomy stent was difficult to reach the target position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Success rate of immediate recanalization | Within 24 hours post-procedure
  The criteria for successful immediate recanalization were target recanalization with a mTICI grade of 2b or 3 grade

SECONDARY OUTCOMES:
mRS 0-2 ratio | pre-procedure, and 90 days post-procedure
  The ratio of mRS 0-2 points = the number of subjects with mRS 0-2 points 90 days after surgery/the number of subjects receiving thrombectomy by intracranial thrombectomy device ×100%
The time from femoral artery puncture to vascular recanalization or the end time of surgery for patients with no vascular recanalization | intra-operative
  Vascular recanalization time = successful recanalization time - femoral artery puncture time
The NIHSS score decreased the rate of subjects with > 4 points | pre-procedure, 24 hours and 7 days post-procedure
  The ratio of subjects with NIHSS score decreased > 4 points = the number of subjects with NIHSS score decreased > 4 points/the number of subjects with thrombotic stent thrombectomy ×100% in this group
Success rate of instrument operation | intra-operative
  Device operation success = the number of devices completed conveying, releasing and retracting in the group/the number of all test devices used in the group ×100%
The incidence of symptomatic intracranial hemorrhage within 24 h post-procedure | within 24 hours post-procedure
  Symptomatic intracranial hemorrhage within 24 h, specifically intracranial hemorrhage (intracranial parenchymal hematoma, subarachnoid hemorrhage, and ventricular hemorrhage) accompanied by neurological deterioration (NIHSS score increased by ≥4 points compared with preoperative)
Mortality within 90 days | within 90 days
  All-cause mortality = the number of deaths in this group/the number of subjects receiving intracranial thrombectomy stent for thrombectomy in this group ×100%
Incidence of device defects | intra-operative
  Defects of research devices during clinical trials, such as broken devices, incorrect labeling, etc
Incidence of SAE (serious adverse events) | intra-operative, 24 hours, 7 days and 90 days post-procedure
  Incidence of SAE = number of subjects with SAE/number of subjects receiving thrombectomy with intracranial thrombectomy device ×100%
Incidence of AE (adverse events) | intra-operative, 24 hours, 7 days and 90 days post-procedure
  Incidence of AE = number of subjects with AE/number of subjects receiving thrombectomy with intracranial thrombectomy device ×100%

CONTACTS AND LOCATIONS:
Overall Officials: Xinfeng Liu, Principal Investigator — General Hospital of Eastern Theater Command, PLA
Locations (1):
- General Hospital of Eastern Theater Command, PLA, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huo S, Gao J, Lv Q, Xie M, Wang H, Zhang X, Xie Y, Wu M, Liu R, Liu X, Yuan K, Ye R. Trajectories of stroke severity and functional outcomes after endovascular treatment in ischemic stroke: A post hoc analysis of a randomized controlled trial. Clin Neurol Neurosurg. 2024 Apr;239:108248. doi: 10.1016/j.clineuro.2024.108248. Epub 2024 Mar 16. PMID 38507987